CLINICAL TRIAL: NCT02940028
Title: ICU Experience Among Family Members of ICU Patients
Brief Title: ICU Experience in Family Members
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1050308
Record Dates: First submitted 2016-10-12; First posted 2016-10-20 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Post-Traumatic Growth, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive writing intervention (Experimental): The intervention group will participate in a brief expressive writing intervention.
  Interventions: Behavioral: Expressive writing
- Control writing intervention (Other): The control group will receive a control writing condition (fact based writing).
  Interventions: Behavioral: Control writing

INTERVENTIONS:
Behavioral: Expressive writing — Brief expressive writing intervention
  Arms: Expressive writing intervention
Behavioral: Control writing — Brief fact-based writing exercise.
  Arms: Control writing intervention

SUMMARY:
The ICU is a stressful and challenging place for patients and their families. Many family members experience anxiety, depression, and post-traumatic stress disorder during and after their ICU experience. The investigators are studying post-traumatic growth in this study. Post-traumatic growth (PTG) is a set of positive changes that occurs after a challenging or difficult life experience. This study investigates the effects of expressive writing on positive changes that occur after a difficult experience. PTG will be compared between the intervention group receiving the expressive writing intervention and the control group (non-expressive or fact based writing).

ELIGIBILITY:
Inclusion Criteria:

Family members of ICU patients are eligible for the study. We will enroll one study participant per patient admitted to a study ICU (Shock Trauma or Respiratory ICU at Intermountain Medical Center) who meets the following inclusion criteria:

* Participant can be a family member of a patient admitted to a study ICU for >24 hours and ≥1 of the following:

  * mechanical ventilation via endotracheal tube for ≥ 12 hours
  * non-invasive ventilation (CPAP, BiPAP) for > 4 hours in a 24-hour period provided for acute respiratory failure in an ICU (not for obstructive sleep apnea or other stable use)
  * high flow nasal cannula or face mask O2 with FiO2 ≥ 0.5 for ≥4 hours
  * use of vasopressors for shock of any etiology for >1 hour
* Both participant and ICU patient must be adult (age ≥18 years of age)
* Participant must be able to read, speak, and write in English
* Participant must be enrolled within 72 hours of the patient's meeting mechanical ventilation criteria

Participants who live with the patient will be accorded higher priority than those who do not live with the patient because they are more likely to be involved as caregivers. The preference would be for the participant to be the designated power of attorney; if there is no designated power of attorney living with the patient, then the primary informal caregiver (identified either by the patient or by the family) would be enrolled; if either of these is not available, the default surrogate (defined in figure 1) would be enrolled. If no one living with the patient meets these criteria, then family members and informal caregivers not living with the patient will be screened for the study. The preference would again be for first, the designated power of attorney, then a primary caregiver and a default surrogate. An informal caregiver provides care without reimbursement.

Exclusion Criteria:

* Pregnant or breastfeeding females
* Prisoners
* Children (age <18 years of age)
* Known history of PTSD, dementia, or schizophrenia. Presence of these illnesses will be per participant report of physician diagnosis and treatment
* If a patient has been transferred from another ICU after an ICU course greater than 24 hours, or if the patient has had a previous ICU or long term acute care (LTAC) admission in the last 90 days, the family member or caregiver will be excluded.
* Patients admitted for hospice
* Participants who live more than 200 miles away or who have no specified domicile
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-04-29 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Growth Inventory | 4 months

SECONDARY OUTCOMES:
Hospital Depression and Anxiety Scale | 4 months
Impact of Event Scale Revised (IES-R) | 4 months
Perceived Stress Scale | 4 months
Brief COPE | 4 months
Physical Symptoms Scale | 4 months
Groningen Activity Restriction Scale (GARS) | 4 months
Activity Restriction Scale | 4 months
Essay Evaluation Measure | 4 months
  The essay evaluation measure assesses if the writing sample (essay) was personal, meaningful and reveals emotions. This measure has 3 items that are scored 0 to 6 for a total score of 0 to 18.

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Hopkins, PhD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02940028/Prot_001.pdf